CLINICAL TRIAL: NCT01891565
Title: Stroke Inpatients Rehabilitation With Accelerometer-based Feedback Reinforcement of Activity
Brief Title: Stroke Inpatients Rehabilitation Reinforcement of Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, Dr. Mayowa Owolabi, Consultant Neurologist, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2013-001
Record Dates: First submitted 2013-06-26; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Activity Feedback (Experimental): Feedback
  Interventions: Behavioral: Feedback
- No Feedback (No Intervention)

INTERVENTIONS:
Behavioral: Feedback
  Arms: Activity Feedback

SUMMARY:
The amount of active therapy provided to patients on an inpatient stroke rehabilitation unit has been reported as often insufficient. Observational studies have found that in the first 14 days post stroke, patients receive very little therapy and have very low activity levels. More opportunity to practice may, however, improve short-term outcomes such as the level of mobility, endurance, use of the affected arm and leg, and length of stay. The Stroke Inpatient Rehabilitation Reinforcement of ACTivity (SIRRACT) trial will utilize sensors that reveal the type, quantity, and aspects of quality of patient activities outside of the confines of research laboratories. SIRRACT will deploy inexpensive Personal Activity Monitors (PAMs), comprised of triaxial accelerometers worn on the thighs.

The objectives of the study are:

i. To assess the impact of feedback from Personal Activity Monitors (PAM)s on amount of active practice, walking speed and distance in stroke patients undergoing rehabilitation.

ii. To assess the impact of feedback from PAMs on physical, psycho-emotional, cognitive and ecosocial Health-Related Quality of Life of stroke patients undergoing rehabilitation.

iii. To assess the acceptability of thigh-strapped accelerometer use among stroke patients undergoing rehabilitation.

iv. To assess the reliability and validity of thigh-strapped accelerometer use among stroke patients undergoing rehabilitation.

Hypotheses In moderate to severely disabled subjects who are receiving in-patient rehabilitation, daily feedback from PAMs about purposeful activity will increase the amount of active practice by >30%, a higher proportion of subjects who reach the level of independence for walking, and increase walking speed by 25%, leading to higher mean walking speeds and distances at the time of discharge from inpatient rehabilitation. Daily feedback from PAMs on increase in walking speed and distances will improve physical, psychological, cognitive and ecosocial domains of Health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Admission for acute inpatient neurorehabilitation of a first stroke (or second stroke after full recovery from prior Transient Ischemic Attack/Stroke).
* Time from onset of stroke to admission for rehabilitation <35 days.
* Stroke from any cause (thrombotic infarct, cardioembolism, intracerebral hemorrhage) that includes unilateral hemiparesis. Hemiparesis means less than or equal 4/5 strength by the British Medical Council scale for hip flexion tested supine and for knee or ankle flexion and extension (scores less than or equal 22 of 25)
* Ability to follow simple instructions, especially to understand verbal reinforcement about activity.
* Independent in mobility prior to admission.
* Able to walk with no more than physical assistance of 2 persons for at least 3 meters. Subjects can use any type of assistive device and brace needed.
* Able to understand and repeat information related to the Informed Consent

Exclusion Criteria:

* Current medical disease that will limit physical therapy at the time of randomization or limited walking prior to the stroke, such as serious infection, Deep Vein Thrombosis, orthostatic hypotension, > stage 2 decubitus ulcer of buttocks or legs, congestive heart failure, claudication, and pain with weight-bearing or walking. Subjects can be entered if a complication resolves within 7 days of admission screening.
* Aphasia with inability to follow 2-step directions during therapeutic instructions or answers Yes/No to questions with greater than or equal 75% accuracy related to personal health and symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change in walking speed | Baseline, Two weeks, Discharge, 1 month
Change in Health-Related Quality of Life as measured using HRQOLISP-26 | Baseline, Two weeks, Discharge, 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mayowa O Owolabi, Principal Investigator — University of Ibadan
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria